CLINICAL TRIAL: NCT06447350
Title: Alcohol Consumption: Norms, Identities, & Motivations (ADUC-Volet 3 " Prevention ")
Brief Title: Alcohol Consumption: Norms, Identities, & Motivations
Acronym: ALCONIM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23-0278
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-10

CONDITIONS: Binge Drinking; Alcohol Drinking
Keywords: norms; induced hypocrisy paradigm; identity; social identity mapping; motivation
MeSH Terms: conditions — Binge Drinking; Alcohol Drinking | interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: 1. control condition with motivational interview
  2. IH condition with motivational interview avec IH program
  3. SIM condition with motivational interview avec SIM program
  4. MM condition with motivational interview avec MM program
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- control (MI) (Active Comparator): A motivational Interview will be conducted with participant.
  Interventions: Behavioral: motivational interviewing
- IH (Experimental): motivational Interview + IH task
  Interventions: Behavioral: Induced hypocrisy; Behavioral: motivational interviewing
- SIM (Experimental): motivational Interview + SIM task
  Interventions: Behavioral: social identity mapping; Behavioral: motivational interviewing
- MM (Experimental): motivational Interview + MM task
  Interventions: Behavioral: Motivational modeling; Behavioral: motivational interviewing

INTERVENTIONS:
Behavioral: Induced hypocrisy — Induced hypocrisy task
  Arms: IH
Behavioral: social identity mapping — Social identity mapping task
  Arms: SIM
Behavioral: Motivational modeling — Motivational modeling task
  Arms: MM
Behavioral: motivational interviewing — motivational interviewing

SUMMARY:
The emergence of new problematic alcohol consumption practices among young people requires new dynamics in prevention strategies. In this context, the ADUC project (Alcohol and Drugs at the University of Caen) aims to develop a better understanding of alcohol consumption, and in particular the practice of binge drinking (BD), in order to develop relevant and adapted prevention tools. The ALCONIM study (IRESP funding; Agreement 20II31-00 - ADUC part 3) is a randomized controlled trial that focuses on the specific determinants of norms, identities and motivations. The main objective of this experiment in social psychology is to validate a program for the prevention of BD practices based on motivational interviewing (MI) associated with induced hypocrisy (IH), social identity mapping (SIM) and motivational modeling (MM) in a student environment.

DETAILED DESCRIPTION:
Context. The emergence of new problematic alcohol consumption practices among young people requires new dynamics in prevention strategies. In this context, the ADUC project (Alcohol and Drugs at the University of Caen) aims to develop a better understanding of alcohol consumption, and in particular the practice of binge drinking (BD), in order to develop relevant and adapted prevention tools. The first step, logistically supported by the University of Caen, consisted in identifying the levels of alcohol consumption of students, the prevalence of binge drinking, and their determinants. Based on more than 7000 participants interviewed, it essentially demonstrated 1) an alarming 22% prevalence of BD among students and 2) three main psychological determinants (see Mange et al., 2021), namely subjective norm (i.e., perception of what is done and/or approved by peers), drinker identity (i.e., how the individual defines him/herself as a drinker), and motivations to drink (social, compliance, enhancement, or coping motivations). Objective. The ALCOMEDIIT study (IRESP funding; Agreement 20II31-00

- ADUC part 3) is a randomized controlled trial . The main objective of this experiment in social psychology is to validate three programs for the prevention of BD practices based on motivational interviewing (MI) associated either induced hypocrisy (IH), social identity mapping (SIM) and motivational modeling (MM) in a student environment..

Materials and Methods. This study will include 240 healthy subjects who will be students at the University of Caen Normandy. They will be people who consume alcohol, having a BD score > 1 in the month preceding the inclusion but not presenting any specific disorder. The trial will be proposed to them by e-mail and the people who meet the inclusion criteria will join either a control group which will benefit from a MI, or an experimental group which will also benefit from a MI but which will be associated with one out of our three psycho-social interventions (IH vs. SIm vs. MM). In order to measure the effectiveness of each prevention program in terms of reducing the use of BD, a follow-up at 1 month (T1) as well as a follow-up at 6 months (T6; exploratory) will be proposed to all participants. The total duration of this research protocol is almost two years. Hypothesis tested. The aim of this work is to evaluate the interest of associating IH, SIM or MM with a motivational interview in a prevention program aiming at reducing alcohol use and the practice of BD in the student population.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 and 30 years old,
* of French mother language,
* of both sexes,
* binge drinking score > 1,
* having signed an informed consent.

Exclusion Criteria:

* Pregnant or breastfeeding students,
* students who declare a history of neurological, neurosurgical, psychiatric, endocrine or infectious diseases.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-04-05 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Binge drinking score | 1 month
  The BD score is calculated on the basis of 3 distinct elements (Q1: "number of average standard drinks per hour (containing about 10g of pure alcohol in France)"; Q2: "number of drunken episodes in the last month" and Q3; "percentage of drunken episodes among the occasions of drinking"). The score results from the following weighting: (4 x Q1) + Q2*6 + (0.2 x Q3). This score considers both the quantity and frequency of drinking, thus integrating the dimension of repeated alcohol withdrawal.

SECONDARY OUTCOMES:
craving | 1 month
  1 item measuring craving
craving | 6 months
  1 item measuring craving
Readiness to Change Alcohol consumption | 1 month
  This self-assessment based on the transtheoretical model of behaviour change (Prochaska & DiClemente, 1982, DiClemente & Prochaska, 1982) is recognized for its reliability and validity. The RTC-Alcohol has three different scales that correspond to an assessment of the three main stages of behaviour change: the pre-contemplation, contemplation and action stages. Based on the person's score on each of these scales, the experimenter determines which stage of behavior change the person is in.
Readiness to Change Alcohol consumption | 6 months
  This self-assessment based on the transtheoretical model of behaviour change (Prochaska & DiClemente, 1982, DiClemente & Prochaska, 1982) is recognized for its reliability and validity. The RTC-Alcohol has three different scales that correspond to an assessment of the three main stages of behaviour change: the pre-contemplation, contemplation and action stages. Based on the person's score on each of these scales, the experimenter determines which stage of behavior change the person is in.
alcohol use | 1 month
  number of alcoholic drinks
alcohol use | 6 months
  number of alcoholic drinks
Binge drinking score | 6 months
  The BD score (Townshend & Duka, 2005) is calculated on the basis of 3 distinct elements (Q1: "number of average standard drinks per hour (containing about 10g of pure alcohol in France)"; Q2: "number of drunken episodes in the last 6 months" and Q3; "percentage of drunken episodes among the occasions of drinking"). The score results from the following weighting: (4 x Q1) + Q2 + (0.2 x Q3). This score considers both the quantity and frequency of drinking, thus integrating the dimension of repeated alcohol withdrawal.
Norm measure | 1 month
  The "Norm measure" questionnaire assesses the "social norm" perceived by participants, i.e., the extent to which a person perceives that those close to him/her approve of and/or practice excessive alcohol consumption. Participants are asked to indicate their degree of agreement on six Likert scales ranging from 1 = strongly disagree to 7 = strongly agree51 , giving a single score based on the average of responses to the 6 items.
Norm measure | 6 months
  The "Norm measure" questionnaire assesses the "social norm" perceived by participants, i.e., the extent to which a person perceives that those close to him/her approve of and/or practice excessive alcohol consumption. Participants are asked to indicate their degree of agreement on six Likert scales ranging from 1 = strongly disagree to 7 = strongly agree51 , giving a single score based on the average of responses to the 6 items.
Alcohol Self-concept Scale | 1 month
  The Alcohol Self-concept Scale (ASCS) assesses the extent to which excessive drinking is important in defining a person's identity. Participants are asked to indicate their level of agreement on five Likert scales, ranging from 1 = strongly disagree to 7 = strongly agree, which will result in a single score based on their averages.
Alcohol Self-concept Scale | 6 months
  The Alcohol Self-concept Scale (ASCS) assesses the extent to which excessive drinking is important in defining a person's identity. Participants are asked to indicate their level of agreement on five Likert scales, ranging from 1 = strongly disagree to 7 = strongly agree, which will result in a single score based on their averages.
Drinking motives questionnaire | 1 month
  The Drinking Motives Questionnaire Revised distinguishes 4 types of drinking motivation: social, coping, enhancement and compliance. These dimensions are evaluated on 12 scales ranging from 1 = never to 5 = always.
Drinking motives questionnaire | 6 months
  The Drinking Motives Questionnaire Revised distinguishes 4 types of drinking motivation: social, coping, enhancement and compliance. These dimensions are evaluated on 12 scales ranging from 1 = never to 5 = always.

CONTACTS AND LOCATIONS:
Locations (1):
- CAEN University Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: No
Study protocol and statistical analysis plan will be shared

REFERENCES:
- [Derived] Lehoux T, Cabe N, Dupont MA, Fleury M, Hamonniere T, Lemercier-Dugarin M, Mauduy M, Mauny N, Montcharmont C, Mortier A, Senemeaud C, Mange J. ALCOhol use, Norms, Identities and Motivations-based (ALCONIM) prevention program for binge drinking among college students: a study protocol for a parallel-group randomized controlled trial. Trials. 2025 Dec 5;27(1):25. doi: 10.1186/s13063-025-09272-0. PMID 41345666